CLINICAL TRIAL: NCT05835817
Title: Magnetoencephalography by Optical Pumping Magnetometer
Acronym: MEG OPM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PI2021_843_0205
Record Dates: First submitted 2023-04-13; First posted 2023-04-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Magnetoencephalography; Optical Pump Magnetometer; Neonate; Premature
Keywords: Magnetoencephalography; optical pump magnetometer; neonate; Premature
MeSH Terms: conditions — Premature Birth | interventions — Magnetoencephalography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adults (Experimental)
  Interventions: Other: Magnetoencephalography
- full term neonates (Experimental)
  Interventions: Other: Magnetoencephalography
- premature neonates (Experimental)
  Interventions: Other: Magnetoencephalography
- pregnant women (Experimental)
  Interventions: Other: Magnetoencephalography

INTERVENTIONS:
Other: Magnetoencephalography — 40 minutes of Magnetoencephalography with Optical Pump Magnetometer

SUMMARY:
MagnetoEncephaloGraphy (MEG) is a method of recording brain activity with high temporal resolution and good spatial resolution, compared to current recording techniques such as ElectroEncephaloGraphy (EEG). The main limitation of MEG is its cost due to the sensors used, the Super Quantum Interference Devices (SQUID). These require a complex infrastructure from an instrumentation point of view to operate, requiring liquid helium, most often at a loss, at increasing cost. Optical Pumping Magnetometers (OPM) type sensors represent a promising alternative to SQUIDs sensors, especially since they do not require helium cooling.

The purpose of this project is to Identify biomarkers in Magnetoencephalography of normal brain development in healthy adults, premature and term newborns from "a priori" obtained by the classical technique of High Resolution EEG performed.

ELIGIBILITY:
Inclusion Criteria:

* For healthy adult volunteers
* Age between 18 and 65
* No pathology, no treatment
* No toxicant intake
* For term newborns
* Child between 38 and 42 weeks gestational age on the day of registration
* No pathology, no treatment
* For children born prematurely
* Child between 28 and 36 weeks gestational age on the day of registration
* No pathology, no treatment apart from routine care related to prematurity
* For pregnant women
* Pregnant with between 28 to 40 weeks gestational age on the day of registration
* No pathology, no treatment

Exclusion Criteria:

* Subject and Patients "not compatible" MEG. Wearers of prosthesis or pacemaker likely to generate artefacts interfering with the measurement. There is no danger to the subject, but the measurement itself may be impossible.
* Patients who cannot stand to stand still for a few minutes.
* Newborn on ventilatory assistance or infusion
* Newborn baby not meeting the age criteria

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Signal to noise ratio of the MEG OPM | 1 day
  Signal to noise ratio of the MEG OPM is in dB
Signal to noise ratio of HR EEG | 1 day
  Signal to noise ratio of HR EEG is in dB
Number of dB between Signal to noise ratio of the MEG OPM and Signal to noise ratio of HR EEG | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No